CLINICAL TRIAL: NCT01969604
Title: Reduction of Daily Sitting Time in Patients With Rheumatoid Arthritis. A Randomized Controlled Trial.
Brief Title: Reduction of Daily Sitting Time in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Tanja Thomsen, PhD-student, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JR-Sedentary Behaviour
Record Dates: First submitted 2013-10-17; First posted 2013-10-25 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Sedentary Behaviour; Motivational Counselling; Short Text Message Service; Fatigue; Pain; Self-efficacy; ActivPAL
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational lifestyle counselling (Experimental): This arm will include 1) Three individual motivational counselling sessions including handouts of four key messages regarding reduction of daily sitting time in combination with 2) Individual Short Text Message (SMS) reminders.
  Interventions: Behavioral: Motivational Lifestyle Counselling
- Control Group (No Intervention): A control group will be encouraged to maintain their usual lifestyle during the 16-week intervention period.

INTERVENTIONS:
Behavioral: Motivational Lifestyle Counselling — The intervention will focus on individual goal setting and self-efficacy, where participants describe their everyday life in terms of sitting time and set goals how to reduce their daily sitting time. Project staff will introduce the patients to the possible benefits of reducing their daily sitting time.
  The intervention focuses on 4 key messages or themes, which are written in booklets that will be handed to the patients: 1) Reduce daily TV-viewing, 2) Substitute sitting with standing when possible, 3) Break up prolonged sitting and 4) Maximum 30 minutes of sitting.
  Based on the patients' own individually goals the patients decide how many weekly SMS reminders they want to receive during the 16-week intervention period.Example:
  • Hello X. Raise from your table stand-up and allow gravity to assist your lunch to digest. Bonus: You burn more energy when you stand.
  Arms: Motivational lifestyle counselling

SUMMARY:
Background:

In recent years there has been a growing interest in sedentary behaviour defined as activities performed in sitting or lying position during waking hours. Sedentary behaviour has been recognised as an independent risk factor for cardiovascular diseases and mortality. A few intervention studies in older sedentary people and in overweight or obese adults have demonstrated, that daily sitting time can be reduced through behavioural intervention.

Patients with rheumatoid arthritis (RA) have an increased risk for cardiovascular diseases, partly caused by the rheumatic disease itself but also because of physical inactivity. Studies have documented a positive effect of increasing physical activity on pain and physical functioning in patients with RA. However, the studies also show, that the patients find it difficult to maintain the increased physical activity levels over time. Previous studies suggest that in promoting health among patients with mobility disability should not solely focus on increasing moderate to vigorous physical activity but also target reduction of sedentary behaviour and increase of light physical activity. In the present study we will focus on reduction of daily sitting time and increase of light physical activity as this approach may prove more feasible for patients with RA.

Objectives and hypothesises:

We hypothesise, that sedentary behaviour can be reduced in patients with RA through a behavioural lifestyle change. In addition, we hypothesize, that reduction of daily sitting time can have a positive effect on symptoms and general health in patients with RA.

The primary objective of the present intervention study is to investigate the effect of a motivational counselling intervention on daily sitting time in adult men and women with RA. Furthermore we want to investigate whether a reduction in daily sitting time is related to reduction in pain and fatigue, reduced weight and waist circumference and improved quality of life, physical function and improved cardiovascular biomarker levels (cholesterol and blood pressure).

Study setting and allocation:

In total, 150 participants will be recruited from the rheumatology outpatient clinic at Glostrup University Hospital, Denmark. The participants will be allocated to either an intervention group (75) or a control group (75).

Intervention:

The intervention aims to support and strengthen the participants' belief in their own ability to reduce their daily sitting time. The intervention will include 1) three individual motivational counselling sessions (60-90 minutes), conducted by one of four project nurses in combination with 2)Individual Short Text Messages (SMS). The counselling sessions will focus on information about the positive health effects of reducing daily sitting time and the participants' own goals of reducing their sitting time. Based on the goals the participants will receive weekly SMS reminders.

Data collection:

Measurements on all participants will be done four times during 22 months; 1) at baseline, 2) 16 weeks after start (by the end of the intervention), 3) six months after end of intervention and 4) 18 months after end of intervention. At each of the four visits the participants fill in questionnaires regarding demographics, lifestyle, daily sitting time, physical activity, physical function, pain , fatigue and quality of life. Furthermore, two occupational therapists will measure the participants' blood pressure, height, weight and waist circumference. At the same time a little monitor will be placed on the participants' thigh, which they will carry for seven days. The monitor measures the participants' physical activity level. The four measurements also include a blood sample from the participants in order to measure cholesterol levels.

DETAILED DESCRIPTION:
Background and rationale:

Physical inactivity is an established risk factor for chronic disease and premature death. In addition to physical inactivity sedentary behaviour has been recognised as a distinct and independent risk factor for cardio metabolic morbidity and mortality in an increasing number of population-based observational studies. Patients with rheumatoid arthritis (RA) have an increased risk for cardio metabolic disease and pre-mature death. The increased risk is, partly caused by the chronic autoimmune rheumatic disease itself and partly to traditional risk factors e.g. hyperlipidemia and hypertension, but can also be attributed to physical inactivity. In Denmark 67 % of patients with RA do not comply with public health recommendations for daily moderate and vigorous physical activity (MVPA), and equivalent proportions are found in Germany (68 %) and the United Kingdom (67 %). Everyday life of patients suffering from RA is periodically influenced by high disease activity (flares) with symptoms such as swelling and stiffness of the joints accompanied by intense pain, leading to severe limitations in physical functioning and potential progressive joint destruction. Intervention studies in patients with RA have documented a positive effect of exercise on pain and physical functioning. However, studies have also demonstrated that exercise and increased activity levels are difficult to maintain over time. Pain has been identified as a main barrier against adaptation and maintenance of a physically activity lifestyle.

Sedentary behaviour can be defined as low metabolic cost activities performed in sitting or reclining positions during waking hours. Sedentary behaviour has become increasingly prevalent in modern society, and recent population studies using self-reported questionnaires estimate daily sitting time of 8-9 hours per day, corresponding to 50-60 % of waking hours in adult general population samples. Likewise, an American population-based study among 4.757 adults, found an objectively measured daily sitting time of 8.44 hours. A few studies have monitored objectively measured sitting time in patients with chronic disease and mobility disability, and these studies generally find that higher proportions of the day are spent sitting among people with various types of mobility disability, i.e. stroke (86-88 % of waking hours), multiple sclerosis (75-85 % of waking hours) and Parkinson's disease (76 % of waking hours). However, to our knowledge no studies have reported objectively measured sitting time in patients with RA. A review from 2011 suggests that aiming to increase PA levels among patients with mobility disability should not solely focus on increasing MVPA, but should also target reduction of sedentary time and increase of light intensity activity, as this approach may prove feasible for improving health and well-being among sedentary patients with chronic disease and mobility limitation.

A few short term intervention studies in older people, and in overweight or obese adults have demonstrated that sedentary behaviour can be reduced through behavioural intervention and that physical activity energy expenditure may be increased by reduction of TV-viewing time. All studies applied objective measures of sitting time.

Objectives:

We hypothesize that sedentary behaviour can be reduced in patients with RA through behavioural lifestyle change. The primary objective of the present randomised trial is to investigate the effect of an individually tailored, theory-based motivational counselling intervention on daily sitting time in patients with rheumatoid arthritis and with sitting time more than 5 hours a day. The secondary objectives are to explore whether a reduction in daily sitting time is related to reduction in pain and fatigue, improved health-related quality of life (HRQOL), self-reported physical function and self-efficacy and improved cardiovascular biomarker levels, and to assess the cost-effectiveness of the intervention.

Design:

The 'Joint Resources' sedentary behaviour intervention study (JR-Sedentary Behaviour) is a randomised, controlled, observer-blinded trial with two parallel groups and a primary endpoint of changes in objectively measured daily sitting time.

Study setting:

Patients will be recruited from lists of patients with RA from the rheumatology outpatient clinic at Copenhagen University Hospital, Glostrup, the Capital Region of Denmark (approximately 2000 patients annually).

Recruitment, screening and participants:

The patients' medical records will be screened for diagnosis code and the latest HAQ-score. Potentially eligible patients will receive a letter with an invitation together with written information about the study and a folder with basic information about trials and personal rights in accordance with the guidelines of the Danish Scientific Ethical Committees. A few days later the daily project leader will call them and ask about their interest in participating in the study. If they are interested they must answer two "screening questions" on 1) self-reported daily sitting time during leisure and work, and 2) self-reported participation in vigorous physical activity (both questions are from The Physical Activity Scale (PAS 2.1)). If eligible the patients will be invited to an information session with the project leader. It will be possible for the patients to sign the consent form immediately following the session or alternatively during the following two days.

Sample size:

Calculation of sample size was based on data from a completed feasibility study (publication under preparation) in which the total daily time in patients with RA was objectively measured with ActivePAL. The daily average sitting time was 10.13±1.7 hours (mean±SD). In the present intervention study we expect a reduction in average daily sitting time of 50 minutes in the intervention group. This estimate is based on an American pilot study from 2012 on obese office workers who reduced their daily sitting time by 48 minutes as a result of the intervention. Based on results from that study, a significance level α = 5%, and a power of 80% we need to include 62 patients in each of the groups. To compensate for attrition we aim to recruit 75 patients in each group.

Randomization and blinding:

Immediately following the baseline measurements randomization to either (A) intervention group (N = 75) or (B) control group (N = 75 ) will be performed via computer-generated "random numbers" for each of the two groups (blocks of 10 patients). Patients will be informed by the project leader about their group allocation one week after baseline measurements. All measurements are conducted by two occupational therapists who will be blinded to group allocation.

Intervention:

The intervention will include 1) Individual motivational counselling including handouts of four key messages regarding in reduction of daily sitting time in combination with 2) Individual Short Text Message (SMS) reminders.

1. Individual motivational counselling The intervention consists of three individual motivational counselling (60-90 minutes) sessions, conducted by one of four nurses or occupational therapists, who are trained to conduct this specific intervention. The first counselling will take place immediately after randomization and allocation to the intervention group, the second counselling two weeks after, and the third counselling ten weeks after the first counselling.

   Contents of motivational counselling The intervention will focus on individual goal setting and self-efficacy, where participants describe their everyday life in terms of sitting time and decide how to reduce their daily sitting time, how to overcome barriers and what goal, in terms of reducing sitting time, they aim for. Motivational counselling techniques will be used.

   First, project staff will introduce the patients to the possible benefits of reducing their daily sitting time. Secondly, project staff will ask the patients to describe their typical day in order to identify resources and barriers for reduction of daily sitting time and discuss possible solutions to overcome barriers and use resources. Thirdly, the patients set their own goals for reduction of daily sitting time using a "catalogue of ideas", which contains proposals to reduce and create breaks in sitting time. Specific proposals to reduce daily sitting time are for example to stand up during phone conversations or TV-watching, get up frequently to go to the printer, get up at least once every half hour and walk around, get up to change the TV channel, make one cup of coffee each time. During the motivational counselling session number two and three patients own goals will be evaluated, new goals will be set and possible solution strategies will be addressed. The patients' motivation and confidence in their own ability to change will be in focus in the last two sessions.

   The intervention program focuses on 4 key messages or themes, including ideas and suggestions for reduction of sitting time, which are written in booklets that will be handed to the patients at each session. The four key messages are: 1) Reduce daily TV-viewing, 2) Substitute sitting with standing when possible - at work and/or at home, 3) Break up prolonged sitting - by standing up frequently and 4) Maximum 30 minutes of sitting per episode.
2. Individual SMS reminders

Based on the patients' own individually goals the patients decide how many weekly SMS reminders they want to receive during the 16-week intervention period and at what time of the day. Examples of SMS text messages are shown below:

* Hello X. Raise from your table stand-up and allow gravity to assist your lunch to digest. Bonus: You burn more energy when you stand.
* Hi X. Regard vacuum cleaning as a free fitness hour. Put music in your ears and do not stop until both the list and the cleaning is done.
* Hi X. You have some truly privileged colleagues who in this afternoon will be able to see you stand by your table. Show them how to do it, and they might follow your good example.
* Hey X. Put the remote control next to the TV if you turn on the television today. Every time you change the channel your entire body gets some exercise.

Control group:

The control group will be encouraged to maintain their usual lifestyle during the 16-week intervention period.

Participant timeline:

The trial will last 22 months including a 16-week intervention and an 18 months follow-up.

Data collection:

Measurements will be done four times during the 22 months 1) at baseline; 2) by end of the intervention (16 weeks after intervention start); 3) six months after the intervention ends and finally (4) 18 months after the intervention ends. At each time patients fill in self-complete questionnaires regarding demographics, lifestyle, sitting time at work and in leisure time, physical activity, physical function, pain, fatigue, health-related quality of life (HRQoL) and self-efficacy. Subsequently, blood pressure, height, weight, waist circumference are measured by two occupational therapists. Blood sampling tests will be taken at Department of Diagnostics, Division of Clinical Biochemistry, Copenhagen University Hospital, Glostrup and store the tests. Baseline demographic characteristics of patients are collected via self-reported questionnaire (using iPad). The two occupational therapists also put on an ActivPAL monitor, which objectively measures the participants' physical activity level for a period of seven days. One week (7 days) after baseline measurements the participant will return to the hospital for removal of the ActivPAL. At the same time they will be informed by TT about the group allocation. One week after each of the follow up measurement the patients will return the ActivPAL in a closed envelope. During each 7 day-period with ActivPal the patients fill in a diary about their non-wear-and sleep time in order to isolate their sitting time from non-wear and sleeping. The patients will be recruited from the DANBIO database, a nationwide registry that has included > 25,000 patients with inflammatory arthritis in a longitudinal observational cohort. At each medical visit in the outpatient clinic, the treating rheumatologist registers information in DANBIO including data regarding disease characteristics (e.g. patient-reported outcomes, disease activity, functional status, disease course) and medical treatment.

Data management:

Since all data will be supplied directly by the patients and the assessors through an online interface via an iPad, there is no risk of data loss or data distortion along the way. Data will be stored encrypted and in unidentifiable form (using participant-numbers) in the server at Glostrup Hospital. Standard missing data analysis will determine if unexpected missing data due to participant drop-out are random or not.

Analysis:

Descriptive statistics and regression analyzes will be conducted. Data analyses will be based on intention-to-treat principle . The scoring of the standardized questionnaires will be made according to the guidelines from instrument developers.

A cost analysis will report the resource use and cost of the intervention. For both the intervention and control group survey and registry based data on resource use including services provided in the health care sector (primary and secondary care) and pharmaceuticals will be aggregated for each individual in intervals determined by the time of data collection. Cost data will be interpolated to total cost for the whole observation period (18 months). The aggregated cost data will be analyzed as costs attributable to the intervention (i.e. difference in difference) and reported as mean values with 95% (bootstrap) confidence intervals. Due to the non-normal distribution of cost data generalized linear models will be employed with appropriate choice of link function.

The analysis of cost-effectiveness will compare the observed gain in QALY (HRQOL over 18 months) with the observed incremental cost (over 18 months) by estimating incremental cost-effectiveness ratios (ICER). To express statistical uncertainty in the ICER estimates acceptability curves will be developed to express the likelihood of the intervention being cost-effective at various QALY threshold values.

The regression model will allow controlling for the baseline value of the study endpoints and other confounding variables that may impact changes in sedentary behavior (e.g. age, gender). In addition, a drop-out analysis will be conducted. Treatment outcomes will be examined using mixed effect models, Bonferroni-correcting for multiple comparisons. All analysis will be carried out with SAS statistical software 9.3.

Ethics, confidentiality and dissemination:

The trial will be performed in accordance with the Helsinki Declaration. The project has been reviewed by the Regional Committee on Biomedical Research Ethics September 2012 as registry based research. The study was approved by the Danish Data Protection Agency. All formal rules and safety rules in the process from data collected for publication are observed (Danish Data Protection Agency, Research Ethics Committee, Clinicaltrial.gov, IT issues, etc.). Anyone who has access to the full relevant data sets (Chief Executive, all supervisors, project staff) are familiar with the formal and safety rules. All information collected during the course of the study will be kept strictly confidential in accordance with Danish Data Protection Agency rules; operationally, this will include consent from the patients.

It is planned to publish at least four scientific papers in peer reviewed journals based on the trial .

In addition, following sources are included in the communication plan:

* Papers (scientific and popular science)
* Presentations at conferences or similar (International and National)
* Collaboration with The Danish Rheumatism Association both members and groups of employees

Access to data:

The project group will have access to data as well as DanBio . Data generated in the trial belong to Copenhagen University Hospital, Glostrup. The steering group to "Joint Resources" will be involved in the case of query about access to data.

Trial status:

Recruitment for the trial is planned to start in April 2013, and will end in December 2014.

Funding:

The study is supported by grants from the Danish Rheumatism Association, the Novo Nordic Foundation, the Lundbeck Foundation, the Research Foundation of the Capital Region of Denmark, the Bevica Foundation, Maersk McKinney Møller Foundation, the Tryg Foundation (external scientific review process), Glostrup Hospital, and Capital Region of Denmark. The funders had no role in the design or management of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA (defined by the American College Rheumatology (ACR) criteria)
* Over the age of 18 years
* Self-reported sitting time for five hours or more per day (measured by Physical Activity Scale, PAS 2.1)
* Physical function score <2.5 (measured by Health Assessment Questionnaire, HAQ)
* Informed consent
* Understand and speak Danish
* Access to mobile phone.

Exclusion Criteria:

* Severe physical disabilities (HAQ-score > 2.5) which would prevent them from reducing daily sitting time (e.g. use of wheelchair);
* Pregnancy
* Vigorous physical activity for more than eight hours a week (measured by PAS 2,1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Changes in daily sitting time in hours and minutes | Baseline, 4 months, 10 months and 22 months
  Changes in objectively measured daily sitting time will be obtained using an ActivPAL® Activity Monitor. This is a small and light uniaxial accelerometer-based device that is worn anteriorly on the upper right thigh and kept in place by waterproof dressing and adhesive tape. The monitor uses accelerometer-derived information about thigh position to estimate time spent in different body positions (i.e. sitting/lying, standing and walking). The activPAL monitor is currently considered the best choice for objective measurement of sitting/lying.
  Changes in self-reported sitting time at work and during leisure time will be measured by the Physical Activity Scale 2.1 (PAS 2.1), a modified version of the original PAS questionnaire, which has previously been validated against accelerometry, PA logs and maximum oxygen uptake. Respondents are asked to specify number of hours and minutes on an average 24-hour day spent on sitting at work and during leisure time.

SECONDARY OUTCOMES:
Fatigue | Baseline, 4 months, 10 months and 22 months
  The 20-item Multi-dimensional Fatigue Inventory (MFI 20) will be included to measure fatigue. MFI 20 consists of 20 statements such as "I feel enthusiastic" and classifies fatigues in five dimensions: 1) General fatigue 2) Physical fatigue 3) Mental fatigue 4) Reduced activity 5) Reduced motivation.
Pain | Baseline, 4 months, 10 months and 22 months
  The Visual Analogue Scale (VAS) transforms the subjective experience of pain to a measurable size. The participant indicates his or her pain by putting a mark on the line where the ends are marked with "no pain" to "worst imaginable pain".
Physical Function | Baseline, 4 months, 10 months and 22 months
  Health Assessment Questionnaire (HAQ) is an instrument that contains 20 questions with four possible answers in eight categories of functions within the ADL (regular daily activities): dressing, rising, eating, walking, personal hygiene, to stretch for something, grab objects and everyday activities. In addition, the HAQ includes VAS scales pain, fatigue and general health.
Health Related Quality of Life (HR-QOL) | Baseline, 4 months, 10 months and 22 months
  HR-QOL is assessed with 1) SF-36, which is a generic instrument consisting of 36 items divided into eight scales: physical function, role physical activity limitations, pain, general health, vitality, social function, role emotional activity limitations and mental health and 2) EuroQol (EQ-5D-5L), which is a standardized 5 item-instrument developed in order to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5 L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Self-efficacy | Baseline, 4 months, 10 months and 22 months
  The General Self-Efficacy Scale assesses a general sense of perceived self-efficacy with the aim to predict coping with daily hassles and adaptation after experiencing stressful life events. The instrument is a 10-item scale with statements such as "I can usually handle whatever comes my way" and "I am confident that I could deal efficiently with unexpected events". The response format is 'not at all true', 'hardly true', 'moderately true', 'exactly true'. The instrument is translated and validated for Danish conditions.
Anthropometric measures | Baseline, 4 months, 10 months and 22 months
  Weight is measured in light clothing without shoes to the nearest 0.1 kg; waist circumference is measured midway between the lower rib margin and the iliac crest to the nearest 0.5 centimetre, without any pressure to the skin and with an unstretched tape meter; hip circumference is measured at the point yielding the maximum circumference over the buttocks to the nearest 0.5 centimetre. The tape should be held in a horizontal plane touching the skin but not indenting the soft tissue. Body mass index (BMI, kg/m2) and waist-hip ratio are calculated.
Blood pressure | Baseline, 4 months, 10 months and 22 months
  Blood pressure will be measured three times at the right upper arm (average of the three measurements) with the participant is in a sitting/lying position; rest 5-10 minutes before the measurements.
Serum Lipids | Baseline, 4 months, 10 months and 22 months
  Venous blood sample will be drawn (not fasting). Total cholesterol, high-density lipoprotein cholesterol (HDL), and triglycerides will be measured by an enzymatic method on the Vitros 5.1 FS from Ortho Clinical Diagnostics. Low-density lipoprotein cholesterol (LDL) and very low-density lipoprotein cholesterol (VLDL) will be calculated by the following formulae (VLDL=Triglyceride x 0.45; LDL=Total cholesterol - HDL + VLDL). Furthermore, C-reactive protein (CRP) and HbA1c will be measured on Vitros 5.1 FS and G8 HPLC Analyzer from TOSOH.

OTHER OUTCOMES:
Cost data | Baseline, 22 months
  For the analysis of intervention costs patients-related activities will be registered for each individual patient by the health care providers. In addition, data will be collected on time use related to each activity and relevant unit cost of resources. Other resource use and cost related to health care provisions will be obtained for each individual patient from the national health registries for hospitals, primary care and purchase of prescription medication from primary care pharmacies. These data will be obtained from the National Board of Health.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Al Esbensen, Research Manager, Principal Investigator — Research Unit of Nursing and Health Science, Glostrup University Hospital, Copenhagen
Locations (1):
- Research Unit of Nursing and Health Science, Glostrup University Hospital, Copenhagen, Denmark, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Sorensen J, Esbensen BA, Aadahl M, Hetland ML, Thomsen T. Cost-effectiveness of motivational counselling and text reminders in patients with rheumatoid arthritis: results based on a randomised clinical trial. RMD Open. 2022 Jul;8(2):e002304. doi: 10.1136/rmdopen-2022-002304. PMID 35853676
- [Derived] Thomsen T, Aadahl M, Beyer N, Hetland ML, Loppenthin KB, Midtgaard J, Christensen R, Nielsen SM, Ostergaard M, Jennum P, Esbensen BA. Sustained Long-Term Efficacy of Motivational Counseling and Text Message Reminders on Daily Sitting Time in Patients With Rheumatoid Arthritis: Long-Term Follow-up of a Randomized, Parallel-Group Trial. Arthritis Care Res (Hoboken). 2020 Nov;72(11):1560-1570. doi: 10.1002/acr.24060. PMID 31507095
- [Derived] Thomsen T, Aadahl M, Beyer N, Hetland ML, Loppenthin K, Midtgaard J, Christensen R, Ostergaard M, Jennum PJ, Esbensen BA. The efficacy of motivational counselling and SMS reminders on daily sitting time in patients with rheumatoid arthritis: a randomised controlled trial. Ann Rheum Dis. 2017 Sep;76(9):1603-1606. doi: 10.1136/annrheumdis-2016-210953. Epub 2017 Jun 5. PMID 28584189
- [Derived] Thomsen T, Aadahl M, Beyer N, Hetland ML, Loppenthin K, Midtgaard J, Christensen R, Esbensen BA. Motivational counselling and SMS-reminders for reduction of daily sitting time in patients with rheumatoid arthritis: a descriptive randomised controlled feasibility study. BMC Musculoskelet Disord. 2016 Oct 18;17(1):434. doi: 10.1186/s12891-016-1266-6. PMID 27756265
- [Derived] Esbensen BA, Thomsen T, Hetland ML, Beyer N, Midtgaard J, Loppenthin K, Jennum P, Ostergaard M, Sorensen J, Christensen R, Aadahl M. The efficacy of motivational counseling and SMS-reminders on daily sitting time in patients with rheumatoid arthritis: protocol for a randomized controlled trial. Trials. 2015 Jan 27;16:23. doi: 10.1186/s13063-014-0540-x. PMID 25623388